CLINICAL TRIAL: NCT04633330
Title: Evaluation of Efficacy of AHCC®for the Clearance of High Risk-HPV Infections in Chinese Female: A Multi-centre, Randomised, Double Blind and Placebo-controlled Study
Brief Title: Evaluation of AHCC® for the Clearance of High Risk-HPV Infections in Chinese Female
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Beihua Kong, Professor, PhD, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHCC-WM-0520
Record Dates: First submitted 2020-10-26; First posted 2020-11-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: High Risk Human Papillomavirus Infection; Low Grade Squamous Intraepithelial Lesion
Keywords: HR-HPV; AHCC®
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): AHCC®capsules, 5 capsules * 3 times per day, empty stomach (defined as one hour before meal or two hours after meal).
  Interventions: Drug: AHCC®capsules
- Control Arm (Placebo Comparator): Simulation of AHCC®capsules, 5 capsules * 3 times per day, empty stomach (defined as one hour before meal or two hours after meal).
  Interventions: Drug: Simulation of AHCC®capsules

INTERVENTIONS:
Drug: AHCC®capsules — AHCC®capsules, a standardized extract of cultured Lentinula edodes mycelia (ECLM) TID for 6 months after enrolment.
  Other Names: Yinuojin Ruanjiaonang
  Arms: Study Arm
Drug: Simulation of AHCC®capsules — TID for 6 months after enrolment. A compensation of AHCC®is provided to participant from control arm when HR-HPV positive at 6 months after enrolment.
  Other Names: Yinuojin Ruanjiaonang Moniji
  Arms: Control Arm

SUMMARY:
This is a multi-centre, randomised, double blind, placebo-controlled study on female participants with diagnosis of high-risk human papillomavirus (HR-HPV) infection to evaluate the clearance capacity of AHCC®.

DETAILED DESCRIPTION:
Worldwide, cervical cancer is the fourth most common malignancy in women and a major cause of morbidity and mortality. It accounts for nearly 10% of all cancers. The etiology of cervical cancer has been identified and confirmed associated with high risk-human papillomavirus (HR-HPV). When HR-HPV infections persist overtime, patients have an increased risk of developing cervical cancer The proprietary, a standardized extract of cultured Lentinula edodes mycelia (ECLM), AHCC®, was developed in Japan in 1992. Several studies have reported a variety of therapeutic effects, including antioxidant and anticancer activity and improvement of immune response.

As recently reported study on AHCC®, pre-clinical in vitro and in vivo evidence demonstrated its durable clearance of HR-HPV infections. The preliminary data from the two pilot studies suggested that AHCC® supplementation supports the host immune system for successful clearance of HR-HPV infections. A confirmatory phase II randomized, double-blinded, placebo-controlled study is about completion. The preliminary results of this phase II study confirmed data observed in pilot studies that AHCC® supplementation for at least 6 months is associated with a 60% successful elimination of HPV infections and confirmed IFN-β correlates with clearance of persistent HPV infections. The optimal duration of AHCC® supplementation required after the first negative result still needs more evaluation in future clinical studies.

Nevertheless, all above mentioned studies have included western participants solely. The aim of this study is to evaluate the clearance capacity of AHCC® on Chinese female participants with diagnosis of HR-HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form
* Not menopausal
* Met persistent HR-HPV infection criteria:
* At least one HR-HPV positive test over 12 months prior to screening
* HR-HPV positive diagnosis by Cobas assay within 3 months prior to screening
* Low grade squamous intraepithelial lesion (LSIL) diagnosis by cytology within 6 months prior to screening
* Willing to take effective contraception method during study period.
* Negative urine pregnancy test within 7 days prior to screening
* Normal haematology, kidney and liver functions: ANC≥1,500 cells/mm3, platelets 100,000≥cells/mm3, creatinine clearance ≥60mL/min (estimated using Cockcroft Gault equation), total bilirubin, serum alanine aminotransferase (SGPT), serum aspartate aminotransferase (SGOT), and alkaline phosphatase ≤ normal value 1.5 Times.

Exclusion Criteria:

* With following medical history within 6 months prior to screening: myocardial infarction, unstable angina, heart failure, or un-controlled hypertension (>140/90 mmHg)
* Systemic treatment for HR-HPV infection has been performed within three months before screening
* Acute genital tract infection
* Previously or currently diagnosed as malignant tumour
* The cytological diagnosis is: ASC-H, AGC tends to become tumorous and other high-risk lesions
* The histological diagnosis is High grade squamous intraepithelial lesion (HSIL)
* Pregnant or breastfeeding
* A history of hepatitis (autoimmune, A, B, or C) or positive antigen
* There is a clear history of mental confusion (schizophrenia, two-way affection, psychosis) or uncontrolled epilepsy
* The main gynaecologist believes that there are significant medical complications, including immunosuppressive conditions (such as HIV, Rheumatoid arthritis, etc.) or are taking immunomodulators (such as immunosuppressive agents)
* Participants with autoimmune diseases
* Taking AHCC® capsules before screening
* Taking other immune-modulating nutritional supplements
* Planned hysterectomy (excluding subtotal hysterectomy)
* Considered by investigators as unsuitable participant of this study

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
High risk human papillomavirus (HR-HPV) infection testing, ROCHE, Cobas assay | 6 months for all participants since enrolment
  The Cobas human papillomavirus (HPV) test is NMPA-approved for cervical and endocervical samples collected in PreservCyt (ThinPrep) media. The Cobas HPV test detects DNA of the high-risk types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68. This test does not detect DNA of HPV low-risk types (e.g., 6, 11, 42, 43, 44) since these are not associated with cervical cancer and its precursor lesions.

SECONDARY OUTCOMES:
Interferon Beta Test-Plasma | 3 months and 6 months for all participants since enrolment, extra-6 month for responding participant from study arm, extra 3 months and 6 months for compensated participants from control arm.
  Human IFN-β (Interferon beta) ELISA Kit will be applied for this test. This kit was based on sandwich enzyme-linked immune-sorbent assay technology. Capture antibody was precoated onto 96-well plates. And the biotin conjugated antibody was used as detection antibodies. The standards, test samples and biotin conjugated detection antibody were added to the wells subsequently, and washed with wash buffer. HRP-Streptavidin was added and unbound conjugates were washed away with wash buffer. TMB substrates were used to visualize HRP enzymatic reaction. TMB was catalysed by HRP to produce a blue colour product that changed into yellow after adding acidic stop solution. The density of yellow is proportional to the target amount of sample captured in plate. Read the O.D. absorbance at 450nm in a microplate reader, and then the concentration of target can be calculated.

OTHER OUTCOMES:
Liquid based cytology test | 6 months for all participants since enrolment, extra-6 month for responding participant from study arm, and extra 6 months for compensated participants from control arm.
  In this method, the cervical cells are immersed in a conserving liquid before being fixed on the slide, avoiding desiccation and reducing the quantity of obscuring material. Liquid cytology can be prepared by manual or automated methods, and various systems are commercially available. They are mostly used for cervical cancer screening but are also adapted for FNAC samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
The desensitised protocol and metadata will be publicly available after completion.
Supporting Information: Study Protocol
Time Frame: The sharing data will be available after Dec. 2021.